CLINICAL TRIAL: NCT04192656
Title: The Effect of Positive Airway Pressure on Idiopathic Sudden Sensorineural Hearing Loss Comorbided With Obstructive Sleep Apnea: A Clinical Randomized Controlled Study
Brief Title: The Effect of PAP on ISSHL Comorbided With OSA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Principal Investigator, Ye Jingying, Director of the dept. of Otolaryngology, Head and Neck Surgery, and Director of the Center of Sleep Medicine, Beijing Tsinghua Chang Gung Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BTCHENT201901
Record Dates: First submitted 2019-12-09; First posted 2019-12-10 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Sudden Hearing Loss; Obstructive Sleep Apnea
MeSH Terms: conditions — Hearing Loss, Sudden; Sleep Apnea, Obstructive | interventions — Methylprednisolone Hemisuccinate; Methylprednisolone; ginaton; Ginkgo biloba extract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PAP plus medication (Experimental): patients treated by both PAP and medication
  Interventions: Device: non-invasive positive airway pressure; Drug: Methylprednisolone Hemisuccinate; Drug: Ginaton
- medication (Active Comparator): patients treated by medication only
  Interventions: Drug: Methylprednisolone Hemisuccinate; Drug: Ginaton

INTERVENTIONS:
Device: non-invasive positive airway pressure — non-invasive positive airway pressure is the first-line treatment for obstructive sleep apnea
  Arms: PAP plus medication
Drug: Methylprednisolone Hemisuccinate — Methylprednisolone is the first-line treatment of idiopathic sudden sensorineural hearing loss
  Other Names: Methylprednisolone, MP
Drug: Ginaton — ginnaton is ginkgo biloba extract
  Other Names: Ginkgo biloba extract,GBE

SUMMARY:
This clinical randomized controlled study is to explore the effect of positive airway pressure(PAP) on patients in Beijing Tsinghua Changgung Hospital diagnosed with both idiopathic sudden sensorineural hearing loss comorbided(ISSHL) and obstructive sleep apnea(OSA) between Dec. 2019 to Dec. 2029.

ELIGIBILITY:
Inclusion Criteria:

1. aged >= 18 and <= 70,
2. diagnosed with OSA by full-night in-lab or home-stay PSG according to AASM 2012 criteria, and AHI > 15/h,
3. diagnosed with ISSHL by AAO-HNS 2019 criteria,
4. ISSHL onset within 1 week.

Exclusion Criteria:

1. sudden hearing loss with certain causes,
2. with severe comorbid diseases,
3. pregnant or breast-feeding women,
4. AHI <= 15/h,
5. hearing threshold recovered > 50% when included,
6. previously regularly treated with PAP.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
hearing threshold | 3 months after onset of ISSHL
  the recovery of hearing threshold which will be measured by pure tone audiometry

CONTACTS AND LOCATIONS:
Overall Officials: Juanjuan Gao, MD, Principal Investigator — Beijing Tsinghua Changung Hospital; jingying Ye, MD, Study Chair — Beijing Tsinghua Changung Hospital; Haijin Yi, MD, Study Director — Beijing Tsinghua Changung Hospital; Mu He, MD, Principal Investigator — Beijing Tsinghua Changung Hospital; Xin Cao, MA, Principal Investigator — Beijing Tsinghua Changung Hospital; Xingxing Lu, MA, Principal Investigator — Beijing Tsinghua Changung Hospital; Sichao Liang, MA, Principal Investigator — Beijing Tsinghua Changung Hospital
Locations (1):
- Beijing Tsinhgua Changgung Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Hizli O, Ozcan M, Unal A. Evaluation of comorbidities in patients with OSAS and simple snoring. ScientificWorldJournal. 2013 Apr 18;2013:709292. doi: 10.1155/2013/709292. Print 2013. PMID 23710145
- [Background] Kayabasi S, Iriz A, Cayonu M, Cengiz B, Acar A, Boynuegri S, Mujdeci B, Eryilmaz A. Vestibular functions were found to be impaired in patients with moderate-to-severe obstructive sleep apnea. Laryngoscope. 2015 May;125(5):1244-8. doi: 10.1002/lary.25021. Epub 2014 Nov 12. PMID 25388224
- [Background] Casale M, Vesperini E, Potena M, Pappacena M, Bressi F, Baptista PJ, Salvinelli F. Is obstructive sleep apnea syndrome a risk factor for auditory pathway? Sleep Breath. 2012 Jun;16(2):413-7. doi: 10.1007/s11325-011-0517-x. Epub 2011 Apr 9. PMID 21479758
- [Background] Fu Q, Wang T, Liang Y, Lin Y, Zhao X, Wan J, Fan S. Auditory Deficits in Patients With Mild and Moderate Obstructive Sleep Apnea Syndrome: A Speech Syllable Evoked Auditory Brainstem Response Study. Clin Exp Otorhinolaryngol. 2019 Feb;12(1):58-65. doi: 10.21053/ceo.2018.00017. Epub 2018 Aug 24. PMID 30134647
- [Background] Sheu JJ, Wu CS, Lin HC. Association between obstructive sleep apnea and sudden sensorineural hearing loss: a population-based case-control study. Arch Otolaryngol Head Neck Surg. 2012 Jan;138(1):55-9. doi: 10.1001/archoto.2011.227. PMID 22249630